CLINICAL TRIAL: NCT01014325
Title: Safety and Efficacy Study With Allergen Extracts of House Dust Mites for Specific Sublingual Immunotherapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Roxall Medizin (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SLG-2009-006B
Record Dates: First submitted 2009-11-11; First posted 2009-11-16 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Allergens

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Allergen extract (Experimental)
  Interventions: Biological: Allergen extract
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Allergen extract — sublingual application
  Arms: Allergen extract
Biological: Placebo — sublingual application
  Arms: Placebo

SUMMARY:
The objective of this clinical trial is to assess the safety and efficacy of sublingual application of allergen extracts for specific immunotherapy in patients suffering from perennial allergic rhinitis due to house dust mites.

ELIGIBILITY:
Inclusion Criteria:

* Positive history of perennial allergic rhinitis
* Positive screening skin prick test (wheal diameter > 3 mm)
* Compliance and ability of the patient to complete a Diary Card for self-evaluating of the symptoms and antisymptomatic medication
* Signed and dated patient´s Informed Consent,

Exclusion Criteria:

* Previous immunotherapy with allergen extracts within the last 3 years,
* Simultaneous participation in other clinical trials,
* Other reasons contra-indicating an inclusion into the trial according to the investigator´s estimation (e.g. poor compliance),
* Auto-immune disorders,
* Severe chronic inflammatory diseases,
* Malignancy,
* Alcohol abuse,
* Existing or intended pregnancy, lactation and/or lack of adequate contraceptive protection,
* Treatment with beta-blockers (incl. local application) and/or other contra-indicated drugs.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Symptom and medication score | 1 year

SECONDARY OUTCOMES:
Safety of sublingual application | 1 year
Protocol of adverse events | 1 year
Quality of Life Questionnaire | 1 year
Evaluation of patients' related clinical global improvement | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Madrid, Spain